CLINICAL TRIAL: NCT05957367
Title: A Master Protocol for the Multi-Cohort, Phase 1/2 Study of DCC-3116 in Combination With Anticancer Therapies in Participants With Advanced Malignancies
Brief Title: A Study of Inlexisertib (DCC-3116) in Combination With Anticancer Therapies in Participants With Advanced Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Deciphera Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DCC-3116-01-002; 2024-516476-15-00 (EU CTIS Number)
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-10

CONDITIONS: GIST
Keywords: Advanced gastrointestinal stromal tumors; gastrointestinal stromal tumors; ripretinib
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — ripretinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation (Part 1, Module A) (Experimental): Escalation Module A Part 1 inlexisertib combination closed on January 8, 2024, with no participants enrolled.
  Interventions: Drug: Inlexisertib
- Expansion (Part 2, Module A) (Experimental): Expansion Module A Part 2 inlexisertib combination closed on January 8, 2024, with no participants enrolled.
  Interventions: Drug: Inlexisertib
- Dose Escalation (Part 1, Module B) (Experimental): Inlexisertib tablets in escalating dose cohorts in 28-day cycles will be administered in combination with ripretinib once daily (QD).
  Interventions: Drug: Inlexisertib; Drug: Ripretinib
- Expansion (Part 2, Module B) (Experimental): Inlexisertib tablets will be administered in combination with ripretinib in 28-day cycles to evaluate preliminary efficacy in participants with 2nd-line advanced gastrointestinal stromal tumor (GIST).
  Interventions: Drug: Inlexisertib; Drug: Ripretinib

INTERVENTIONS:
Drug: Inlexisertib — Oral Tablet Formulation
  Other Names: DCC-3116
Drug: Ripretinib — Oral Tablet Formulation
  Other Names: QINLOCK, DCC-2618
  Arms: Dose Escalation (Part 1, Module B); Expansion (Part 2, Module B)

SUMMARY:
This is a Phase 1/2, multicenter, open-label (unless otherwise specified in a combination-specific module) study of inlexisertib in combination with anticancer therapies. Modules within the master protocol are defined according to different combinations of inlexisertib with other anticancer agents.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age
* Module A: Part 1 and Part 2:

Module A Part 1 and Part 2 inlexisertib combination closed on January 8, 2024, with no participants enrolled.

* Module B: Only for Part 1 (Safety/Dose-finding):

  * Pathologically confirmed diagnosis of GIST with a KIT or platelet-derived growth factor receptor alpha (PDGFRA) mutation
  * Must have progressed on at least one approved systemic regimen given in the locally advanced or metastatic setting or have documented intolerance to it
  * Must not have received prior ripretinib treatment
* Module B: Only for Part 2 (Expansion)

  * Pathologically confirmed GIST with documented mutation in KIT exon 11
  * Must have progressed on imatinib given in the locally advanced or metastatic setting or have been intolerant to imatinib and may not have received additional systemic therapy for GIST
* Must have at least 1 measurable lesion according to Modified Response Evaluation Criteria in Solid Tumors (mRECIST)
* Must have a life expectancy of more than 3 months and an ECOG performance status of 0-1
* Adequate organ function and bone marrow reserve based on laboratory assessments performed at Screening
* Must provide a fresh tumor biopsy, if able

Exclusion Criteria:

* Must not have received the following within the specified time periods prior to the first dose of study drug:

  1. Medications, including anticancer therapies, that are known strong or moderate inhibitors or inducers of CYP3A4 or P-glycoprotein (P-gp) including certain herbal medications (eg, St. John's wort): 14 days or 5×the half-life of the medication (whichever is longer)
  2. Other anticancer therapies and any investigational therapies with a known safety and PK profile: 14 days or 5×the half-life of the medication (whichever is shorter)
  3. Investigational therapies with unknown safety and PK profile: 28 days. If there is enough data on the investigational therapy to assess the risk for drug-drug interactions and late toxicities of prior therapy as low, the Sponsor's Medical Monitor may approve a shorter washout of 14 days
  4. Grapefruit or grapefruit juice: 14 days
* Have not recovered from all clinically relevant toxicities from prior therapy
* New York Heart Association Class III or IV heart disease, active ischemia, or any other uncontrolled cardiac condition, clinically significant cardiac arrhythmia requiring therapy, uncontrolled hypertension, congestive heart failure, or myocardial infarction within 6 months prior to the first dose of study drug
* Symptomatic central nervous system (CNS) metastases or presence of leptomeningeal disease
* Malabsorption syndrome
* Radiation for indications other than bone disease must have been completed 4 weeks prior to first dose of study drug, unless it consisted of limited field palliative radiation, including whole brain radiation, which must have been completed at least 2 weeks prior to first dose of study drug
* Major surgery within 4 weeks of the first dose of study drug
* Active HIV, Hepatitis B or Hepatitis C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (Escalation Phase) | Approximately 24 months
  Identify the observed adverse events and serious adverse events associated with inlexisertib in combination with other anticancer therapies.
Recommended Phase 2 Doses (RP2D) (Escalation Phase) | Approximately 18 months
  Identify the dose-limiting toxicities for each dose level tested and determine the recommended Phase 2 doses of inlexisertib in combination with other anticancer therapies.
Objective response rate (ORR) (Expansion Phase) | Approximately 24 months
  Proportion of participants who achieve CR or PR per histology-specific consensus response criteria.

SECONDARY OUTCOMES:
Duration of response (DoR) | Approximately 24 months
  DoR is defined as the time interval from the time that the measurement criteria are first met for CR or PR (whichever is first recorded) per histology-specific consensus response criteria until the first date that the progressive disease is objectively documented or death, whichever occurs first.
Disease Control Rate (DCR) | Approximately 24 months
  The DCR is defined as the proportion of participants who achieve CR, PR, or stable disease (SD) per histology-specific consensus response criteria.
Time to response | Approximately 24 months
  Time to response is defined as the time from initiation of treatment until the first assessment demonstrating CR or PR per histology-specific consensus response criteria.
Progression-free survival (PFS) | Approximately 24 months
  PFS is defined as the time from initiation of treatment until documented disease progression per histology-specific consensus response criteria or death, whichever occurs first.
Overall Survival (OS) | Approximately 48 months
  OS is defined as the time from initiation of treatment until death.
Maximum observed concentration (Cmax) | Predose and up to 12 hours postdose
  Measure the maximum observed concentration of inlexisertib combinations.
Time to maximum observed concentration (Tmax) | Predose and up to 12 hours postdose
  Measure the time to maximum plasma concentration of inlexisertib combinations.
Minimum observed concentration (Cmin) | Predose and up to 12 hours postdose
  Measure the minimum observed concentration of inlexisertib combinations.
Area under the concentration-time curve (AUC) | Predose and up to 12 hours postdose
  Measure the AUC of inlexisertib combinations.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team, Study Director — Deciphera Pharmaceuticals, LLC
Locations (12):
- United States (11):
  - University of Southern California - Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Department of Medicine-Hematology/Oncology, Los Angeles, California
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Massachusetts Worcester, Worcester, Massachusetts
  - START Midwest, Grand Rapids, Michigan
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center - Main Campus, New York, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Virginia Cancer Specialist, PC, Fairfax, Virginia
- Inselspital Universitätsklinikum Bern, Bern, Switzerland